CLINICAL TRIAL: NCT06418581
Title: Investigation on Burnout of Physicians
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0139
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study proposes to analyze the burnout, emotional states, and sleep conditions of internal medicine doctors at the Second Affiliated Hospital of Zhejiang University School of Medicine through a questionnaire survey. The findings aim to provide reference for implementing measures to address burnout among medical staff, improve their physical and mental health, and enhance the quality of healthcare.

DETAILED DESCRIPTION:
Burnout, proposed by American psychologist Herbert Freudenberger in 1974, is defined as a syndrome resulting from chronic exposure to workplace stressors and the inability to successfully manage them. Subsequently, Maslach et al. considered burnout as the state of emotional exhaustion, depersonalization, and reduced personal accomplishment resulting from prolonged exposure to work-related stressors. In January 2022, the World Health Organization (WHO) included "burn-out" in the 11th Revision of the International Classification of Diseases (ICD-11) for the first time, officially recognizing it as a disease. Burnout is considered a syndrome resulting from chronic workplace stress that has not been successfully managed. Compared to other professions, doctors are at a higher risk of experiencing burnout. Burnout among medical professionals is closely related to job quality, doctor-patient relationships, and overall health. In 2022, 47% of 13,000 physicians in the United States reported experiencing burnout. Investigating whether burnout affects physical and mental health, thereby impacting the quality of healthcare, is essential.

ELIGIBILITY:
Inclusion Criteria:

1. Currently employed or non-employed internists, including those in gastroenterology, cardiology, pulmonology, hematology, rheumatology, endocrinology, general medicine, infectious diseases, oncology, neurology, psychiatry, nutrition, and other related specialties.
2. Ability to complete the questionnaire.
3. No history of mental illness.

Exclusion Criteria:

1. Individuals who are not part of the internal medicine system, such as those in surgery, medical technology departments, or administrative roles.
2. Inability to effectively complete all sections of the questionnaire.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will involve doctors from the internal medicine department of the Second Affiliated Hospital of Zhejiang University who will fill out the survey questionnaire using internet-based methods after providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Investigation and analysis of occupational burnout and psychological status of physicians | 2024.10.1-2025.10.1
  article

CONTACTS AND LOCATIONS:
Overall Officials: Caihua Wang, Doctor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewa CS, Loong D, Bonato S, Trojanowski L. The relationship between physician burnout and quality of healthcare in terms of safety and acceptability: a systematic review. BMJ Open. 2017 Jun 21;7(6):e015141. doi: 10.1136/bmjopen-2016-015141. PMID 28637730
- [Background] Farr E, Lee S, Maltser S, Verduzco-Gutierrez M, Shapiro LT. A rapid response for burnout among inpatient physiatrists: A survey of leaders of inpatient rehabilitation facilities. PM R. 2022 Sep;14(9):1080-1085. doi: 10.1002/pmrj.12870. Epub 2022 Aug 9. PMID 35789206